CLINICAL TRIAL: NCT06656403
Title: Effect of Artificial Tears on Ocular Biometry Parameters
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: He Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IOL2024
Record Dates: First submitted 2024-10-22; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Dry Eye Disease; Tear Film
Keywords: dry eye; IOL Master 700; tear film
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Other): dry eye patients
  Interventions: Drug: 0.1% sodium hyaluronate
- Control group (Other): non-dry eye patients
  Interventions: Drug: 0.1% sodium hyaluronate

INTERVENTIONS:
Drug: 0.1% sodium hyaluronate — After baseline measurement, 0.1% sodium hyaluronate eye drops were instillation into the inferior conjunctival vault of both eyes

SUMMARY:
Due to the instability of the tear film, the biometry often needs to be done multiple times in a clinical environment. The high variability of both short-term and long-term repeatability in keratometry of dry eyes is well-known. Consequently, enhancing the condition of the eye surface in individuals with dry eyes will result in improved precision when choosing the power of intraocular lenses (IOLs). This prospective and before-and-after self-control study will recruit 100 patients.

DETAILED DESCRIPTION:
Over the past ten years, surgery has progressed from rejuvenation surgery to refractive surgery, which focuses on enhancing both vision and addressing pre-existing issues that impact visual quality. This is why good surgical outcomes involve thorough preoperative assessment and precise intraocular lens(IOL) power determination. To achieve the intended postoperative refractive outcomes, it is essential to perform an accurate calculation of intraocular lens power (i.e., biometry), which may impact the accuracy of the computation.

Damage to the eye's surface from chronic inflammation and induced tear film hyperosmolarity occurs in DED because tear film homeostasis is disrupted. The changes in tear film dynamics and damage to the ocular surface result in mistakes in optical measures, which in turn affect the results of procedures like cataract surgery that heavily rely on these assessments.

Consequently, enhancing the condition of the eye surface in individuals with dry eyes will result in improved precision when choosing the power of intraocular lenses (IOLs).

ELIGIBILITY:
Inclusion Criteria:

(1) age ≥18 years,(2) able and willing to comply with the treatment schedule.

Exclusion Criteria:

1. The eyes cannot fixate on the fixation lamp (such as children, nystagmus diseases, severe low vision, inattention, etc.) and cannot act according to the user's instructions and sit in the front of the equipment (the forehead or lower song is injured so that it cannot be supported on the forehead / lower song bracket)
2. The eyes are cloudy with optical media (such as corneal opacity, central corneal scar, mature cataract, posterior chamber bag opacity, vitreous hemorrhage, etc.).
3. The eyelid is completely closed or too small (drooping, relaxation) resulting in complete or partial occlusion of the cornea
4. Just after contact measurement or examination, use a corneal local anesthesia solution. (IOL Master 700 should avoid using local anesthetic before all contact examinations)
5. Tear film deformation (lack of specular reflection of the cornea during corneal curvature measurement), the severity of grade IV dry eye, and whether eye drops were used 24 hours before the examination.
6. Any corneal lesions (corneal irregularity, corneal scar or corrosive burning, severe irregular astigmatism of cornea)
7. Fundus lesions (changes in the anatomical morphology of retinal macular fovea during axial length measurement, such as retinal detachment, edema, ulcer, etc.)
8. Patients with ocular trauma, surgery, and excessive photosensitivity, such as photodynamic therapy (PDT), were excluded.
9. using eye drops (0.1% Sodium hyaluronate) allergic patients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2024-11-20 (Estimated); Study Completion 2024-11-21 (Estimated)

PRIMARY OUTCOMES:
flat meridian of the anterior corneal surface (K1) | Baseline,30s,2min,5min
  K1 was measured using IOL Master 700 for 4 times. To assess the Biometry measurements were assesssed at baseline, 2nd ,3rd and 4th(30-second, 2-minute and 5-minute intervals respectively) time after instilling one drop of ATD (0.1% Sodium hyaluronate, preservative free)
steep meridian of the anterior corneal surface (K2) | Baseline,30s,2min,5min
  K2 was measured using IOL Master 700 for 4 times. To assess the Biometry measurements were assesssed at baseline, 2nd ,3rd and 4th(30-second, 2-minute and 5-minute intervals respectively) time after instilling one drop of ATD (0.1% Sodium hyaluronate, preservative free)
central corneal thickness (CCT) | Baseline,30s,2min,5min
  CCT was measured using IOL Master 700 for 4 times. To assess the Biometry measurements were assesssed at baseline, 2nd ,3rd and 4th(30-second, 2-minute and 5-minute intervals respectively) time after instilling one drop of ATD (0.1% Sodium hyaluronate, preservative free)

SECONDARY OUTCOMES:
axial length (AL) | Baseline,30s,2min,5min
  AL was measured using IOL Master 700 for 4 times. To assess the Biometry measurements were assesssed at baseline, 2nd ,3rd and 4th(30-second, 2-minute and 5-minute intervals respectively) time after instilling one drop of ATD (0.1% Sodium hyaluronate, preservative free)
corneal curvature radius(R1,R2) | Baseline,30s,2min,5min
  R1,R2 was measured using IOL Master 700 for 4 times. To assess the Biometry measurements were assesssed at baseline, 2nd ,3rd and 4th(30-second, 2-minute and 5-minute intervals respectively) time after instilling one drop of ATD (0.1% Sodium hyaluronate, preservative free)
anterior chamber depth (ACD) | Baseline,30s,2min,5min
  ACD was measured using IOL Master 700 for 4 times. To assess the Biometry measurements were assesssed at baseline, 2nd ,3rd and 4th(30-second, 2-minute and 5-minute intervals respectively) time after instilling one drop of ATD (0.1% Sodium hyaluronate, preservative free)
white-to-white corneal diameter (WTW) | Baseline,30s,2min,5min
  WTW was measured using IOL Master 700 for 4 times. To assess the Biometry measurements were assesssed at baseline, 2nd ,3rd and 4th(30-second, 2-minute and 5-minute intervals respectively) time after instilling one drop of ATD (0.1% Sodium hyaluronate, preservative free)
Pupil (Pup) | Baseline,30s,2min,5min
  Pup was measured using IOL Master 700 for 4 times. To assess the Biometry measurements were assesssed at baseline, 2nd ,3rd and 4th(30-second, 2-minute and 5-minute intervals respectively) time after instilling one drop of ATD (0.1% Sodium hyaluronate, preservative free)
non-invasive tear break-up time (NITBUT) | Baseline
  Non-invasive first tear film breakup time using the Keratograph 5M (Oculus, Germany) topographer will be measured three times consecutively and the median value was recorded
tear meniscus height(TMH) | Baseline
  TMH using the Keratograph 5M (Oculus, Germany) topographer will be measured three times consecutively and the median value was recorded
ocular surface disease index(OSDI) | Baseline
  Chinese translated, and validated OSDI (Allergan Inc, Irvine, USA) version will be used to assess and quantify DE symptom. The 12 items of the questionnaire can be tabulated into a score that ranges from 0 (no symptoms) to 100 (severe symptoms) points

CONTACTS AND LOCATIONS:
Overall Officials: Guanghao Qin, Principal Investigator — He Eye Specialist Hospital

REFERENCES:
- [Background] Roggla V, Leydolt C, Schartmuller D, Schwarzenbacher L, Meyer E, Abela-Formanek C, Menapace R. Influence of Artificial Tears on Keratometric Measurements in Cataract Patients. Am J Ophthalmol. 2021 Jan;221:1-8. doi: 10.1016/j.ajo.2020.08.024. Epub 2020 Aug 21. PMID 32828877
- [Background] Nibandhe AS, Donthineni PR. Understanding and Optimizing Ocular Biometry for Cataract Surgery in Dry Eye Disease: A Review. Semin Ophthalmol. 2023 Jan;38(1):24-30. doi: 10.1080/08820538.2022.2112699. Epub 2022 Aug 20. PMID 35989638
- [Background] Chen X, Yuan F, Wu L. Metaanalysis of intraocular lens power calculation after laser refractive surgery in myopic eyes. J Cataract Refract Surg. 2016 Jan;42(1):163-70. doi: 10.1016/j.jcrs.2015.12.005. PMID 26948792
- [Background] Koh S. Irregular Astigmatism and Higher-Order Aberrations in Eyes With Dry Eye Disease. Invest Ophthalmol Vis Sci. 2018 Nov 1;59(14):DES36-DES40. doi: 10.1167/iovs.17-23500. PMID 30481804
- [Background] Koh S, Tung CI, Inoue Y, Jhanji V. Effects of tear film dynamics on quality of vision. Br J Ophthalmol. 2018 Dec;102(12):1615-1620. doi: 10.1136/bjophthalmol-2018-312333. Epub 2018 Jun 15. PMID 29907632
- [Background] Epitropoulos AT, Matossian C, Berdy GJ, Malhotra RP, Potvin R. Effect of tear osmolarity on repeatability of keratometry for cataract surgery planning. J Cataract Refract Surg. 2015 Aug;41(8):1672-7. doi: 10.1016/j.jcrs.2015.01.016. PMID 26432124
- [Background] Sheard R. Optimising biometry for best outcomes in cataract surgery. Eye (Lond). 2014 Feb;28(2):118-25. doi: 10.1038/eye.2013.248. Epub 2013 Dec 6. PMID 24310239
- [Background] Hovanesian J, Epitropoulos A, Donnenfeld ED, Holladay JT. The Effect of Lifitegrast on Refractive Accuracy and Symptoms in Dry Eye Patients Undergoing Cataract Surgery. Clin Ophthalmol. 2020 Sep 16;14:2709-2716. doi: 10.2147/OPTH.S264520. eCollection 2020. PMID 32982163
- [Background] Sahin A, Hamrah P. Clinically relevant biometry. Curr Opin Ophthalmol. 2012 Jan;23(1):47-53. doi: 10.1097/ICU.0b013e32834cd63e. PMID 22081032